CLINICAL TRIAL: NCT05673876
Title: A Phase Ib, Open-label, Randomized, Dose-finding, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of GDC-8264 in Combination With Standard of Care in the Treatment of Acute Graft-versus-Host Disease in Patients Who Have Undergone Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Study to Assess the Safety and Pharmacokinetics of GDC-8264 in Combination With Standard of Care in Participants With Acute Graft-Versus-Host Disease (aGVHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA43861; ISRCTN27200385 (Other: ISRCTN (United Kingdom))
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Acute Graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GDC-8264, 35 mg (Experimental): Participants will receive oral GDC-8264, 35 milligrams (mg), once daily (QD) for 28 days.
  Interventions: Drug: GDC-8264
- GDC-8264, 75 mg (Experimental): Participants will receive oral GDC-8264, 75 mg, PO, QD for 28 days.
  Interventions: Drug: GDC-8264

INTERVENTIONS:
Drug: GDC-8264 — GDC-8264 tablets will be administered as per the schedule specified in the respective arms.

SUMMARY:
The primary purpose of the study is to assess the safety and pharmacokinetics (PK) of GDC-8264 in participants with acute graft-versus-host disease (aGVHD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of post-allogeneic hematopoietic stem cell transplantation (HSCT) aGVHD at screening
* Evidence of engraftment post-transplant
* Diagnosis of high-risk aGVHD, per refined Minnesota high-risk aGVHD criteria during screening
* Initiation of treatment with systemic corticosteroids for aGVHD at a dose of prednisone ≥2 milligrams per kilograms per day (mg/kg/day) by orally (PO) or methylprednisolone ≥2 mg/kg/day intravenously (or equivalent) in divided doses at diagnosis and up to 3 days prior to or on the same day as initiation of GDC-8264 (Day 1), with no taper planned prior to Day 3

Exclusion Criteria:

* Evidence of relapsed, progressing, or persistent malignancy, or treatment for relapse after transplant, or requirement for rapid immune suppression withdrawal as pre-emergent treatment of early malignancy relapse
* Prior receipt of more than one allogeneic HSCT
* Prior receipt of solid organ transplantation that are target organs for aGVHD (e.g., liver transplant)
* Prior systemic treatment for aGVHD, except for the standard of care corticosteroid treatment initiated as part of this trial
* Diagnosis of chronic GVHD or overlap syndrome
* Uncontrolled active infection (i.e., progressive symptoms related to infection despite treatment, or persistently positive blood cultures despite treatment, or any other evidence of severe sepsis)
* Severe organ dysfunction (e.g., acute liver failure, renal failure requiring dialysis, ventilator support, or vasopressor therapy)
* Initiation or planned use of a marketed small molecule (excluding corticosteroids) or biologic therapy as treatment for aGVHD from the start of screening through the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7 participants took part in the study across 4 investigative sites in the United States from 06 April 2023 to 15 January 2024.
Pre-assignment Details: Participants with acute graft-versus-host disease (aGVHD) were randomized in 1:1 ratio to receive GDC-8264, 35 milligrams (mg) or GDC-8264, 75 mg.
Groups:
- GDC-8264 35 mg: Participants received GDC-8264, 35 mg tablets, orally, once daily (QD) in combination with standard-of-care corticosteroid treatment during the 28 day treatment period.
- GDC-8264 75 mg: Participants received GDC-8264, 75 mg tablets, orally, QD in combination with standard-of-care corticosteroid treatment during the 28 day treatment period.
Period: Overall Study
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Started | 4 | 3
Completed | 1 | 0
Not Completed | 3 | 3
Not completed — Death | 3 | 1
Not completed — Study Terminated by Sponsor | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least one dose of GDC-8264, with participants grouped according to treatment received.
Groups:
- GDC-8264 35 mg: Participants received GDC-8264, 35 mg tablets, orally, QD in combination with standard-of-care corticosteroid treatment during the 28 day treatment period.
- Total: Total of all reporting groups
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (12.7) | 57.3 (6.8) | 59.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From signing informed consent form until 28 days after the final dose of GDC-8264 (up to 9 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 4 | 3
Participants | 4 | 3

2. Primary Outcome: Plasma Concentration of GDC-8264
Description: Plasma concentration of GDC-8264 at specified timepoints was determined.
Time Frame: Predose, 1.5, 2, 3, 4, 6, 12, and 24 hours post-dose on Days 1 and 4; Predose on Days 8, 15, 22, 29
Population: Pharmacokinetic (PK) population included participants who received at least one dose of GDC-8264 and had at least one evaluable post-dose PK concentration. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/millilitres (ng/mL)
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 3 | 3
nanograms/millilitres (ng/mL)
  Predose on Day 1: number analyzed (Participants) | 3 | 2
  Predose on Day 1 | NA (NA) — The geometric mean and geometric coefficient of variation was not estimable as the samples were below the limit of quantification (BLQ). | NA (NA) — The geometric mean and geometric coefficient of variation was not estimable as the samples were BLQ.
  1.5 hours Postdose on Day 1: number analyzed (Participants) | 3 | 2
  1.5 hours Postdose on Day 1 | 28.3 (141.5) | 698 (17.0)
  2 hours Postdose on Day 1: number analyzed (Participants) | 1 | 2
  2 hours Postdose on Day 1 | 151 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated. | 835 (10.3)
  3 hours Postdose on Day 1: number analyzed (Participants) | 2 | 2
  3 hours Postdose on Day 1 | 89.7 (321.6) | 858 (57.2)
  4 hours Postdose on Day 1: number analyzed (Participants) | 2 | 2
  4 hours Postdose on Day 1 | 123 (141.1) | 781 (33.8)
  6 hours Postdose on Day 1: number analyzed (Participants) | 1 | 2
  6 hours Postdose on Day 1 | 227 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated. | 700 (52.5)
  12 hours Postdose on Day 1: number analyzed (Participants) | 3 | 2
  12 hours Postdose on Day 1 | 24.0 (28439.7) | 361 (106.5)
  24 hours Postdose on Day 1: number analyzed (Participants) | 3 | 2
  24 hours Postdose on Day 1 | 12.2 (5241.5) | 144 (116.0)
  Predose on Day 4 | 58.9 (167.3) | 167 (78.1)
  1.5 hours Postdose on Day 4 | 400 (27.2) | 195 (158.2)
  2 hours Postdose on Day 4 | 529 (31.8) | 218 (181.5)
  3 hours Postdose on Day 4 | 433 (19.2) | 318 (223.3)
  4 hours Postdose on Day 4 | 374 (8.8) | 393 (175.7)
  6 hours Postdose on Day 4 | 274 (6.7) | 539 (127.1)
  12 hours Postdose on Day 4: number analyzed (Participants) | 2 | 3
  12 hours Postdose on Day 4 | 129 (43.1) | 373 (82.6)
  24 hours Postdose on Day 4 | 43.2 (143.2) | 140 (79.9)
  Predose on Day 8 | 39.5 (138.0) | 266 (70.1)
  Predose on Day 15: number analyzed (Participants) | 2 | 2
  Predose on Day 15 | 6.47 (NA) — Values were less than reportable (LTR) for one participant. Since only one participant was evaluable, the geometric coefficient of variation could not be estimated. | 294 (54.6)
  Predose on Day 22: number analyzed (Participants) | 2 | 2
  Predose on Day 22 | 6.50 (NA) — Values were LTR for one participant. Since only one participant was evaluable, the geometric coefficient of variation could not be estimated. | 276 (180.1)
  Predose on Day 29: number analyzed (Participants) | 2 | 2
  Predose on Day 29 | 61.5 (297.2) | 1.51 (NA) — Values were LTR for one participant. Since only one participant was evaluable, the geometric coefficient of variation could not be estimated.

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of GDC-8264
Description: Steady-state (SS) PK visit was Day 4 if the participant was hospitalized or Day 8 if the participant was an outpatient. If the SS PK visit samples could not be obtained on Day 4/8, the SS PK visit may have occurred on any dosing day between Day 4 and 28.
Time Frame: Day 1 and SS visit (any time between Day 4 to Day 28)
Population: PK population included participants who received at least one dose of GDC-8264 and had at least one evaluable post-dose PK concentration. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 3 | 2
ng/mL
  Day 1: number analyzed (Participants) | 1 | 2
  Day 1 | 270.00 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated. | 991.21 (33.7)
  SS PK Day: number analyzed (Participants) | 3 | 1
  SS PK Day | 541.48 (31.1) | 1480.00 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

4. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of GDC-8264
Description: SS PK visit was Day 4 if the participant was hospitalized or Day 8 if the participant was an outpatient. If the SS PK visit samples could not be obtained on Day 4/8, the SS PK visit may have occurred on any dosing day between Day 4 and 28.
Time Frame: Day 1 and SS visit (any time between Day 4 to Day 28)
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 3 | 2
hours
  Day 1: number analyzed (Participants) | 1 | 2
  Day 1 | 3.4 [3.4 to 3.4] | 2.30 [1.6 to 3.0]
  SS PK Day: number analyzed (Participants) | 3 | 1
  SS PK Day | 2.17 [1.5 to 3.1] | 3.2 [3.2 to 3.2]

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC0-24) of GDC-8264
Description: as for outcome 4
Time Frame: Day 1 and SS visit (any time between Day 4 to Day 28)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/millilitres (ng*hr/mL)
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 3 | 2
nanograms*hours/millilitres (ng*hr/mL)
  Day 1: number analyzed (Participants) | 1 | 2
  Day 1 | 3250.37 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated. | 10528.86 (57.8)
  SS PK Day: number analyzed (Participants) | 3 | 1
  SS PK Day | 4534.44 (24.4) | 19405.83 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

6. Primary Outcome: Terminal Half-life (T1/2) of GDC-8264
Description: as for outcome 4
Time Frame: Day 1 and SS visit (any time between Day 4 to Day 28)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 3 | 2
hours
  Day 1: number analyzed (Participants) | 1 | 2
  Day 1 | 7.03 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated. | 7.82 (27.2)
  SS PK Day: number analyzed (Participants) | 3 | 1
  SS PK Day | 6.84 (50.2) | 8.70 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

7. Primary Outcome: Apparent Clearance (CL/F) of GDC-8264
Description: as for outcome 4
Time Frame: Day 1 and SS visit (any time between Day 4 to Day 28)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millilitres/hours (mL/hr)
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 3 | 2
millilitres/hours (mL/hr)
  Day 1: number analyzed (Participants) | 1 | 2
  Day 1 | 9608.61 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated. | 6131.74 (69.5)
  SS PK Day: number analyzed (Participants) | 3 | 1
  SS PK Day | 6871.73 (32.5) | 3216.19 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

8. Primary Outcome: Apparent Volume of Distribution (Vz/F) of GDC-8264
Description: as for outcome 4
Time Frame: Day 1 and SS visit (any time between Day 4 to Day 28)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millilitres (mL)
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 3 | 2
millilitres (mL)
  Day 1: number analyzed (Participants) | 1 | 2
  Day 1 | 97480.88 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated. | 69212.58 (37.3)
  SS PK Day: number analyzed (Participants) | 3 | 1
  SS PK Day | 67784.28 (21.0) | 40355.80 (NA) — Since only 1 participant was analyzed, geometric coefficient of variation could not be calculated.

9. Secondary Outcome: Overall Response Rate (ORR) on Day 29
Description: ORR=percentage of participants with complete response (CR), very good partial response (VGPR), or partial response (PR) as determined by investigator. CR=all target organs evaluated as Mount Sinai Acute GVHD International Consortium (MAGIC) aGVHD Stage 0 [Skin- no GVHD rash; Liver - bilirubin <2 milligrams/decilitres (mg/dL); Upper gastrointestinal (GI) tract - no intermittent nausea, vomiting/anorexia; Lower GI tract - stool output: < 500 mL/day or <3 episodes/day (adults), <10 mL/kilograms (kg)/day or <4 episodes/day]. VGPR=resolution of signs & symptoms i.e. no rash/residual erythematous rash involving < 25% of body surface, without (w/o) bullae; bilirubin <2 mg/dL or <25% of baseline at screening; toleration of food/enteral feeding; predominantly formed stools; no overt GI bleeding/abdominal cramping; no more than occasional nausea/vomiting. PR=improvement in one/more target organs (skin, liver, upper GI tract, lower GI tract) involved with aGVHD symptoms w/o worsening in others.
Time Frame: Up to Day 29
Population: Modified intent to treat (mITT) included all enrolled participants who received at least one dose of GDC-8264 and did not miss more than four doses of the GDC-8264 within the first 14 days of the treatment period due to participant noncompliance, voluntary withdrawal, or reasons other than safety or (lack of) efficacy. Percentages have been rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 2 | 3
percentage of participants | 100 | 66.7

10. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined astime from response (CR, VGPR or PR) on Day 29 to aGVHD progression from nadir in any organ, new systemic therapy for aGVHD, or death from any cause (whichever occurs first), as determined by the investigator. CR=all target organs evaluated as MAGIC aGVHD Stage 0 [Skin- no GVHD rash; Liver - bilirubin <2 mg/dL; Upper GI tract - no intermittent nausea, vomiting/anorexia; Lower GI tract - stool output: < 500 mL/day or <3 episodes/day (adults), <10 mL/kg/day or <4 episodes/day]. VGPR=resolution of signs & symptoms i.e. no rash or residual erythematous rash involving < 25% of body surface, without bullae; bilirubin <2 mg/dL or <25% of baseline at screening; toleration of food/enteral feeding; predominantly formed stools; no overt GI bleeding or abdominal cramping; no more than occasional nausea or vomiting. PR=improvement in one or more target organs (skin, liver, upper GI tract, lower GI tract) involved with aGVHD symptoms without worsening in others.
Time Frame: From Day 29 up to end of study (up to 9 months)
Population: mITT included all enrolled participants who received at least one dose of GDC-8264 and did not miss more than four doses of the GDC-8264 within the first 14 days of the treatment period due to participant noncompliance, voluntary withdrawal, or reasons other than safety or (lack of) efficacy. Overall number analyzed is the number of participants with OR i.e. responders.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 2 | 2
days | 1.00 [1.0 to 1.0] | 4.00 [4.0 to 4.0]

11. Secondary Outcome: Percentage of Participants With aGVHD Flares by Day 56
Description: aGVHD flare was defined as an increase in aGVHD target organ stage by at least one stage for at least 3 days that requires either addition of a new line of systemic treatment or increase in corticosteroid dose > 0.25 mg/kg/day.
Time Frame: Baseline up to Day 56
Population: mITT included all enrolled participants who received at least one dose of GDC-8264 and did not miss more than four doses of the GDC-8264 within the first 14 days of the treatment period due to participant noncompliance, voluntary withdrawal, or reasons other than safety or (lack of) efficacy. Percentages have been rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 2 | 3
percentage of participants | 50 | 0

12. Secondary Outcome: Percentage of Participants With Non-relapse Mortality (NRM) by Day 180
Description: NRM was defined as any death that occurred after onset of aGVHD that was not attributable to relapse of the underlying primary disease was considered a non-relapse death.
Time Frame: Baseline up to Day 180
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | GDC-8264 35 mg | GDC-8264 75 mg
Number analyzed (Participants) | 2 | 3
percentage of participants | 0 | 66.7

ADVERSE EVENTS:
Time Frame: From signing informed consent form until 28 days after the final dose of GDC-8264 (up to 9 months)
Description: Safety population included participants who received at least one dose of GDC-8264, with participants grouped according to treatment received.
Groups:
- GDC-8264 35mg: Participants received GDC-8264, 35 mg tablets, orally, QD in combination with standard-of-care corticosteroid treatment during the 28 day treatment period.
- GDC-8264 75mg: Participants received GDC-8264, 75 mg tablets, orally, QD in combination with standard-of-care corticosteroid treatment during the 28 day treatment period.
Arm/Group | GDC-8264 35mg | GDC-8264 75mg
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-8264 35mg (N=4) | GDC-8264 75mg (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-8264 35mg (N=4) | GDC-8264 75mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 3 (4) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 2 (3)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT05673876/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT05673876/ICF_001.pdf